CLINICAL TRIAL: NCT01190735
Title: Caffeine for Motor Manifestations of Parkinson's Disease: An Open-Label Dose-Response Study.
Brief Title: Caffeine for Motor Manifestations of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ron Postuma (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Ron Postuma, Neurologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIHR-219243
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
Keywords: Caffeine; Parkinson's Disease; Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases; Caffeine citrate; Molecular Mechanisms of Pharmacological Action; Pharmacologic Actions; Central Nervous System Stimulants; Physiological Effects of Drugs; Central Nervous System Agents; Therapeutic Uses
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caffeine (Experimental): Each patient will take pills twice per day containing 100-200 mg of caffeine (as synthetic caffeine alkaloid). Patients will be instructed to take whatever caffeine-containing beverages they are accustomed to taking, without changing their habitual schedule (note that all will be taking <200 mg per day). Caffeine intake will be assessed at each visit. Patients will continue their usual PD medications, without change in dose or timing for the entire duration of the study. Medication will be provided in pre-packaged dosettes.
  Interventions: Drug: Caffeine alkaloid

INTERVENTIONS:
Drug: Caffeine alkaloid — The following intervention will be provided for six consecutive weeks:
  Week 1 (100 mg BID), Week 2 (200 mg BID), Week 3 (300 mg BID), Week 4 (400 mg BID), Week 5 and 6(500 mg BID). At the conclusion of the study, patients will decrease their dose by 100 mg BID every other day, until caffeine is stopped. This gradual reduction will be to prevent withdrawal symptoms. If a patient experiences a dose-limiting event, they will be terminated from the study, and will withdraw from the medication in the same manner. If dose-limiting events occur between visits, patients will be encouraged to decrease the caffeine dose back to the previously-tolerated dose until in-person assessment can be performed.
  Other Names: Wake-Ups; 100mg tabs, NPN 00533629, serial no 5503701103; 200mg tabs, NPN, 80003474, serial no 5503701105

SUMMARY:
Numerous epidemiological studies have linked lifelong use of caffeine to a lower risk of Parkinson's disease (PD) - prospective studies have estimated that non-coffee drinkers have an approximately 1.7-2.5 fold increased risk of developing PD compared to coffee drinkers. This is an extremely important finding which deserves further more in depth investigations.

The exact pathophysiological mechanism remains elusive, but multiple hypotheses do exist: Caffeine antagonizes adenosine receptors directly yielding an improvement on motor systems and even on Levodopa serum concentrations (when on therapy). An additional explanation is that adenosine antagonism has neuroprotective properties by acting locally on basal ganglia circuits and the substantia nigra.

The current study aims to identify the optimal caffeine dose with maximal motor benefit and the least amount of undesirable adverse effects.

DETAILED DESCRIPTION:
Caffeine has been in widespread use for centuries, and is the commonest psychostimulant used worldwide. In Canada, estimates of mean daily intake for a 70 kg person range from 200-450 mg. The main sources of caffeine ingestion are in beverages - depending on brewing technique a typical cup of drip-filtered coffee can contain between 100 and 150 mg of caffeine (gourmet drip coffees contain up to 300 mg and espresso preparations generally contain much less caffeine). Black tea contains between 30 and 50 mg, and lower amounts of caffeine are found in soft drinks, green teas, and chocolate. Caffeine is a substance with a well-defined effect and side-effect profile, and in general it is very well tolerated. Side effects can include irritability, insomnia, enhancement of physiologic tremor, and stomach upset. Abrupt withdrawal from caffeine can cause headache and excessive sleepiness. Caffeine can exacerbate pre-existing supraventricular tachycardia. Multiple large-scale epidemiologic studies have not found evidence for adverse health effects with long-term moderate use of caffeine. Caffeine has a T-max of approximately 1 hour and readily crosses the blood brain barrier. It has first order kinetics. Plasma half life estimates range from 3-6 hours, increased in the case of pregnancy or severe liver disease. Drug interactions are uncommon: Caffeine withdrawal may cause lithium toxicity, and caffeine increases clozapine levels.

CNS effects of caffeine are mainly due to antagonism of the A1 and A2A adenosine receptors, (A2A predominates in the striatum). Potential effects upon motor manifestations of PD are predominantly related to the antagonistic action of adenosine on dopamine release in the striatum. Partial tolerance to CNS effects is common, and begins to occur within one week (tolerance is more pronounced for the A1 receptor, suggesting that motor changes may show less tolerance). If effective for PD, caffeine has the potential to be a very important advance for patient care, for numerous reasons. First of all, it has been in widespread use for centuries, so the long-term safety has been determined. Caffeine is widely available as tablets which are very inexpensive (i.e. less than 25 cents per tablet), potentially resulting in substantial cost savings for patients and health-care planners. Caffeine also has the potential (as yet unproven) to treat non-motor manifestations of PD, particularly excessive daytime somnolence.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been diagnosed with idiopathic Parkinson's disease (stage I - IV Hoehn and Yahr)

Exclusion Criteria:

1. Estimated daily caffeine intake of more than 200 mg per day.
2. Subject has dementia (MMSE < 26/30) and ADL impairment secondary to cognitive loss, inability to understand consent process.
3. Changes to antiparkinsonian medications in last 4 weeks or changes will be required during the period of the study protocol.
4. Contraindication to caffeine use:

   1. Uncontrolled hypertension (systolic bp >170 or diastolic bp >110 on two consecutive readings)
   2. Use of lithium or clozapine
   3. Pre-menopausal women who are not using effective methods of birth control
   4. Current use of prescribed alerting agents such as modafinil and methylphenidate
   5. Active peptic ulcer disease
   6. Supraventricular cardiac arrhythmia
   7. Previous adverse reaction to caffeine which either required admission to hospital,or after which the patient was directly advised by a physician to not use caffeine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Tolerability | 6 weeks
  Patients will be given a structured questionnaire targeting common side effects of caffeine, as well as a series of open-ended questions for other side effects. Vital signs will be measured. Questionnaire symptoms will be selected, where available, from the common terminology criteria for adverse events, version 3.0, developed by the National Cancer Institute. A severity of 2 or greater on the 5-point scale will delineate a dose-limiting effect. Evaluations will occur in person after 2 weeks, 4 weeks, 6 weeks (at study termination) and via telephone follow-up at the end of weeks 1,3 and 5.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | 6 weeks
  Will systematically track changes in ESS.
Unified Parkinson Disease Rating Scale(UPDRS): Part II | 6 weeks
  Systematically performing part II of the UPDRS, motor examination.
Timed Up and Go (TUG) | 6 weeks
  This is a measure of gait and transfer speed.
Clinical Global Impression of Change | 6 weeks
Pittsburgh Sleep Quality Index | 6 weeks
Fatigue Severity Scale | 6 weeks
The Parkinson's Disease Questionnaire - PDQ-39 | 6 weeks
  This self-completion questionnaire addresses aspects of functioning and well-being in those affected by Parkinson's Disease (PD). Considered to be the industry 'gold standard' in the assessment of quality of life in PD patients. The 39-point PDQ provides scores on 8 scales: mobility, activities of daily living, emotions, stigma, social support, cognition, communications and bodily discomfort.
Beck Depression Inventory | 6 weeks
  Self-administered questionnaire.
Beck Anxiety Inventory | 6 weeks
  Self-administered questionnaire.
UPDRS: Part I,II,IV | 6 weeks
  Systematically querying I (non-motor aspects of activities of daily living), II (motor aspects of activities of daily living) and IV (motor complications)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Postuma, MD, Msc, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre; Robert Altman, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- See also: Ongoing study investigating caffeine for excessive daytime somnolence in Parkinson's Disease — http://clinicaltrials.gov/ct2/show/NCT00459420?term=postuma&rank=1